CLINICAL TRIAL: NCT07008326
Title: Comparative Effects of High-Intensity Circuit Training and Moderate-Intensity Continuous Training on Various Health Parameters in Overweight Young Adults
Brief Title: Comparing HICT and MICT for Health Improvements in Overweight Young Adults
Acronym: HiMod Impact
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Nani Cahyani Sudarsono, Dr. dr. Nani Cahyani Sudarsono, Sp.KO, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-09-1459
Record Dates: First submitted 2025-04-25; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Overweight
Keywords: high intensity circuit training; moderate intensity continuous training; overweight; young adult male
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Circuit Training (Experimental): High Intensity Circuit Training, a bodyweight exercise program performed 3 times per week with increased intensity every 4 weeks
  Interventions: Behavioral: High Intensity Circuit Training
- Moderate Intensity Continuous Training (Active Comparator): Moderate Intensity Continuous Training, brisk walk or jogging based exercise with increased intensity every 2-4 weeks
  Interventions: Behavioral: Moderate Intensity Continuous Training

INTERVENTIONS:
Behavioral: High Intensity Circuit Training — HICT: 3x/week high intensity circuit training for 12 weeks
  Arms: High Intensity Circuit Training
Behavioral: Moderate Intensity Continuous Training — 3x/week moderate intensity continuous training for 12 weeks
  Arms: Moderate Intensity Continuous Training

SUMMARY:
The increasing prevalence of overweight and obesity is becoming a concern worldwide as it is associated with the increased prevalence of non-communicable diseases. One of the main reasons for this problem is that more adults did not fulfill the weekly physical activity recommendations, with the lack of time and motivation as the main factor. This study aims to compare the effectiveness of a high-intensity circuit training program and the more familiar moderate-intensity continuous training in improving body composition, cardiorespiratory fitness, lipid profile, oxidative stress, and inflammatory markers in young adult males. At the same time, it also explores its adherence through its enjoyment scale and gradual changes in supervision. This experimental study compares pre- and post-tests in the two groups. 3-days food records and 7-days physical activity will be measured monthly as the confounding factors.

DETAILED DESCRIPTION:
* Participants will be recruited consecutively via online forms distributed throughout universities and networks across Jakarta and its surrounding area. Interested individuals will go through early screening. Eligible candidates will then complete an initial assessment at the research site.
* Research assistants will use standard operational procedures for each assessment. The training for research assistants will be done before data collection. One group of research assistants are responsible for main outcome data collection. The researcher is responsible for data analysis. Continuous evaluations will be done weekly to improve the research process.
* Sample size is measured from the 6-research outcomes using the sample size calculation formula for evaluating the mean difference between two variables in repeated measurements.
* Eligible candidates who passed the initial assessment will be randomly divided into HICT (intervention) and MICT (control). The 12-week exercise program in both groups will change gradually in volume, intensity, and supervision. Both volume and intensity will be increased according to heart rate targets. Supervision will decrease gradually from fully supervised in the first 4 weeks, partially supervised in the second 4 weeks, and no supervision in the third 4 weeks.
* Data will be collected and electronically recorded during each training session at the research site by the researcher and research assistants. This data includes time, heart rate, blood pressure, rating of perceived exertion (Borg Scale), training intensity, weight used, and enjoyment (PACES).
* Subjects are encouraged to report any problem during intervention via online messaging or during on-site sessions to the research assistants. The reports will be documented in a separate form. The research assistant leading the data collection will ensure that no data is missing by performing daily checking.
* Data collection for the main outcomes will be done by a different group of research assistants and will be masked from the intervention groupings.
* Data analysis will be done using SPSS 26.0 by the researcher. The analysis will be started after baseline measurements are completed. We will present all normally distributed numeric data as mean and standard deviations and non-normally distributed numeric data as median and minimum-maximum range. Bivariate analysis of normally distributed data will be done using repeated 2-way ANOVA test or mixed linear model in case of many dropouts. If data is not distributed normally, the Friedman test will be used. Any missing data will be stated and completed immediately. Close supervision for each subject will be done by research assistance to ensure all necessary reports are collected and analysed.

ELIGIBILITY:
Inclusion Criteria:

* Overweight (BMI 23-24.9 kg/m2)
* Physically inactive in the last 6 months before the study (<150 minutes of moderate-intensity activity and <75 minutes of high-intensity activity)
* Willing to participate in exercise program for 12 weeks
* No other exercise program during the study period

Exclusion Criteria:

* Smoking
* Medical comorbidities (diabetes mellitus, hypertension, cardiovascular disease, asthma, dyslipidaemia, epilepsy)
* History of musculoskeletal injuries or health problems related to exercise in the last 1 year

Dropout Criteria

* Resigning
* Not participating in the endline assessment
* Not participating in the exercise program for 2 consecutive weeks
* Experiencing injury or health problems that led to the inability to participate in the program for 2 consecutive weeks

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index | Week 0, 4, 8, 12
  Weight and Height will be combined to report Body Mass Index in kg/m^2
Body Fat Percentage | Week 0, 4, 8, 12
  The total percentage of body fat mass measured by BIA Tanita MC-780 in %
Muscle Mass | Week 0, 4, 8, 12
  Muscle mass measured by BIA Tanita MC-780 in kilograms
Visceral Fat Mass | Week 0, 4, 8, 12
  Visceral fat mass measured by BIA Tanita MC-780 in kilograms
Waist Circumference | Week 0, 4, 8, 12
  Waist circumference measured in centimeters
Cardiorespiratory Fitness | Week 0, 12
  VO2Max or VO2peak depends on the feasibility. The cardiac output (mL/min) and body weight (kg) will be combined in mL/kg. min
Total Cholesterol | Week 0, 12
  Total cholesterol in blood measured in mg/dL
High-Density Lipoprotein (HDL) | Week 0, 12
  HDL concentration in blood measured in mg/dL
Low-Density Lipoprotein (LDL) | Week 0, 12
  LDL concentration in blood measured in mg/dL
Triglyceride | Week 0, 12
  Triglyceride concentration in blood measured in mg/dL
Superoxide dismutase | Week 0, 12
  Superoxide dismutase concentration in blood from whole blood sample measured in U/mL
Malondialdehyde | Week 0, 12
  Malondialdehyde concentration in blood from whole blood samples measured in micromolar
Tumor Necrosis Factor-alpha | Week 0, 12
  Tumor Necrosis Factor-alpha concentration in blood measured in pg/mL
Interleukin-6 | Week 0, 12
  Interleukin-6 concentration in blood measured in pg/mL

SECONDARY OUTCOMES:
Enjoyment | Up to 12 weeks
  PACES Score results will be between 18 to 126. A higher score indicates a higher enjoyment level.

CONTACTS AND LOCATIONS:
Overall Officials: Nani C Sudarsono, Doctor, Principal Investigator — Fakultas Kedokteran Universitas Indonesia
Locations (1):
- Universitas Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia

REFERENCES:
- [Background] Klika B, Jordan C. High-intensity circuit training using body weight: maximum results with minimal investment. ACSM's Health & Fitness Journal. June 2013; 17(3):p 8-13.